CLINICAL TRIAL: NCT05790187
Title: Face Perception and Impact of Surgical Masks in Preterm Infants
Acronym: Premask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC22.0365
Record Dates: First submitted 2023-02-15; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-01

CONDITIONS: Visual Preference With and Without Mask in Term Infant; Visual Preference With and Without Mask in Preterm Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- visual test (Experimental): Presentation of differents face pictures
  Interventions: Other: Presentation of differents face pictures

INTERVENTIONS:
Other: Presentation of differents face pictures — Test 1: Unmasked face vs. masked face Test 2: Unmasked face up vs. unmasked face down Test 3: Face masked right side vs. face masked reverse

SUMMARY:
The preferences to masked and unmasked faces is relevant for premature newborns, since Covid-19, most of the faces that surround them during their hospitalization are masked. The Premask project is a continuation of the InfantMask and BabyMask studies (concerning infant and newborn), by studying the visual preferences to masked and unmasked faces of premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants born before 32SA arriving at term (at≥37SA) hospitalized in the neonatology department of the pediatric hospital of Grenoble and approaching discharge will be included.

Of the potential participants meeting the inclusion criteria, those with at least 1 of the following exclusion criteria will not be eligible for inclusion in the study.

Exclusion Criteria:

* Parents not fluent in French
* Parents with no social security rights
* Patient with a syndromic disorder
* Abnormal neurological examination Invasive or non-invasive ventilation at the time of testing of babies requiring, at the time of testing at ≥37SA, non-invasive or invasive ventilatory support as well as labeled syndromic or ophthalmologic disease of prematurity (retinopathies).
* Infection requiring isolation
* Ophthalmologic impairment of prematurity (retinopathy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
proportion of visual fixation time to photos of masked/non-masked faces. | once, at term (at 37 weeks corrected age)
  time of picture visual fixation (seconds)

IPD SHARING:
Plan to Share IPD: Undecided